CLINICAL TRIAL: NCT04880343
Title: Randomised, Open-label, Controlled Clinical Trial to Evaluate the Efficacy of a Product Consisting of D Mannose 2 g+ Cran-max 500 mg+ Vitamin D3 0.001 mg (UROMANNOSA®) in Women With Recurrent Lower Urinary Tract Infections
Brief Title: Clinical Study to Evaluate the Efficacy of the Dietary Supplement UROMANNOSA® in Women With Recurrent Lower Urinary Tract Infections
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruiting the control arm in accordance with the protocol prevent the study population from being reached.
Sponsor: Carmen Gonzalez Enguita (Other)
Responsible Party: Sponsor-Investigator, Carmen Gonzalez Enguita, Staff Physician, Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Organization: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FJD-URO-19-001
Record Dates: First submitted 2021-04-29; First posted 2021-05-10 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Lower Urinary Tract Infection
MeSH Terms: interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (C) (No Intervention): Control
- Group (A) (Experimental): Treatment
  Interventions: Dietary Supplement: Group (A)
- Group (B) (Experimental): Treatment
  Interventions: Dietary Supplement: Group (B)

INTERVENTIONS:
Dietary Supplement: Group (A) — Group that will take a daily dose of the commercial dietary supplement provided by the sponsor, composed of mannose, cran-max and vitamin D for 6 months
  Arms: Group (A)
Dietary Supplement: Group (B) — Group that will take a daily dose of the commercial dietary supplement provided by the sponsor, composed of mannose, cran-max and vitamin D for 3 months
  Arms: Group (B)

SUMMARY:
To analyze the clinical impact of a food supplement composed of D Mannose, cranberry extract (Cran-max) and Vitamin D3 in the prevention of recurrent lower urinary tract infections (UTI)

DETAILED DESCRIPTION:
Once patients have been informed about the study, the potential risks and treatment alternatives, those who meet the selection criteria, agree to participate and sign the informed consent, will be randomly and openly assigned, in a 1:1:1 ratio, to one of the following groups:

Group A: Patients with repeat UTIs who will receive prophylactic treatment for 6 Months.

Group B: Patients with repeat UTIs who will receive prophylactic treatment for 3 Months.

Control group: Patients with recurrent UTIs who will not receive as prophylactic treatment the supplement under study.

The three groups will be treated following standard clinical practice with follow-up at 3, 6, 9 and 12 months after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* History of Recurrent Lower Urinary Tract Infection (at least two episodes in the last 6 months or three episodes in the last 12 months).
* Multiple infections must be spaced a minimum of 2 weeks apart or if less, with a negative urine culture in between.
* Women who agree to participate and give their informed consent in writing

Exclusion Criteria:

* Use of antibiotics or cranberry or other preventive treatment, pharmacological or not, for recurrence of urinary tract infections in the last two weeks.
* Patient with indwelling catheter or intermittent catheterization.
* Patients who present: Interstitial Cystitis, Neurogenic Bladder, Diabetes Mellitus, Nephrolithiasis, Cervical-Uterine Cancer diagnosed and treated less than 5 years ago.
* Use of anticoagulants or contraceptive methods using spermicides or diaphragms.
* Women consuming probiotics or foods, beverages or supplements containing extracts or parts of the genus Vaccinum sp, including other forms of V. macrocarpon (blueberry), V. myrtillus (European blueberry), V.angustifolium (wild or lowbush blueberry), V. corymbosum ( highbush blueberry) or V. vitis-ideae (mountain blueberry), during the two weeks prior to recruitment.
* High consumption of fruits rich in phenolic compounds, with special reference to berries.

Women allergic to berries

* Pregnant or breastfeeding women.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Not based on self-representation
Enrollment: 108 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2024-01-26 (Estimated); Study Completion 2024-01-26 (Estimated)

PRIMARY OUTCOMES:
UTI Recurrence | Through study completion, an average of one year
  Number of patients with recurrences (defined as: number of patients with at least one UTI during the study period) at 6 months.
UTI Recurrence | Variable for each participant over course of up to one year
  Time (in days) from the start of treatment to the next episode of UTI
Number of symptomatic UTIs | Variable for each participant over course of up to one year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Fundación Jiménez Díaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No